CLINICAL TRIAL: NCT03253016
Title: A Comparative Evaluation to Evaluate the Correlation Between Cervical Cerclage or Vaginal Progesterone and Maternal Vaginal Microbiome Distribution During Pregnancy
Brief Title: The Impact of Cervical Cerclage or Vaginal Progesterone on Vaginal Microbiome Distribution
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Western Galilee Hospital-Nahariya (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 0196-16-NHR
Record Dates: First submitted 2017-08-14; First posted 2017-08-17 (Actual); Last update posted 2017-08-17 (Actual); Status verified 2017-03

CONDITIONS: Preterm Labor
MeSH Terms: conditions — Obstetric Labor, Premature | interventions — Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- cervicall cerclage (Experimental): to test vaginal microbiome distribution in women with cervical cerclage due to cervical incompetence in weeks: 12 14 18 26 32
  Interventions: Diagnostic Test: vaginal swab -microbiome test and blood test for cytokines
- vaginal progesterone (Experimental): to test vaginal microbiome distribution in women treated with vaginal progesterone due to cervical shortening in weeks: 12 14 18 26 32
  Interventions: Diagnostic Test: vaginal swab -microbiome test and blood test for cytokines
- contol (No Intervention): to test vaginal microbiome during pregnancies without cerclage or progesterone

INTERVENTIONS:
Diagnostic Test: vaginal swab -microbiome test and blood test for cytokines — vaginal microbiome test and blood test for cytokines repeated during pregnancy in the 3 arms
  Arms: cervicall cerclage; vaginal progesterone

SUMMARY:
A comparative evaluation to evaluate the correlation between cervical cerclage or vaginal progesterone and maternal vaginal microbiome distribution during pregnancy

DETAILED DESCRIPTION:
Cervical insufficiency is primarily a clinical diagnosis, characterized by painless cervical dilation leading to recurrent second-trimester pregnancy losses/births of otherwise normal pregnancies.

Adverse perinatal events associated with cervical insufficiency include prolapse of the fetal membranes into the vagina, intra-amniotic infection, preterm premature rupture of membranes, preterm labor and fetal loss.

Congenital and acquired cervical abnormalities increase the risk of cervical insufficiency; Acquired risk factors are more common and include cervical trauma during delivery, rapid mechanical cervical dilation before a gynecologic procedure or treatment of cervical intraepithelial neoplasia (1). Congenital abnormalities include genetic disorders affecting collagen, uterine anomalies and in the past - in utero diethylstilbestrol (DES) exposure (2, 3).

The diagnosis of cervical insufficiency is based on either

* History of painless cervical dilatation with preterm (midtrimester) delivery
* History of prior second-trimester pregnancy losses or preterm births and cervical length ≤25 mm on transvaginal ultrasonography examination or advanced cervical changes on physical examination before 24 weeks of gestation.

The diagnosis of cervical insufficiency is usually limited to singleton gestations. In addition, preterm labor, infection, abruptio placenta, and bleeding placenta previa should be excluded, as these disorders could account for biochemically mediated cervical ripening leading to second-trimester pregnancy loss or preterm delivery independent of structural/anatomic cervical weakness [4].

The American College of Obstetricians and Gynecologists (ACOG) defines cervical insufficiency as the inability of the uterine cervix to retain a pregnancy in the second trimester in the absence of clinical contractions, labor, or both [5].

Women with a history of cervical insufficiency should be considered for history-indicated cerclage in future pregnancies at 12 to 14 weeks of gestation (6, 7).

Cerclage placement is considered a benign proce¬dure, the risks of such procedure include - cervical lacerations at the time of delivery, the need for cesarean delivery because of the inability of the cervix to dilate secondary to cervical scarring and dystocia, infection, cervical cerclage displacement Nonsurgical interventions have been advocated for patients with presumed cervical insufficiency. Progesterone supplementation appears to reduce the rate of spontaneous singleton preterm birth in women who have had a previous spontaneous preterm singleton birth and in women with a short cervix on ultrasound examination in the current pregnancy (8). In women with a prior preterm birth, continuing progesterone supplementation after placement of a cerclage has not been proven to be useful, but available data are limited.

Most cerclages are placed via a transvaginal approach. The transabdominal approach is more invasive, but allows higher placement, while transvaginal cerclages often end up distal to the internal os. The two most common transvaginal techniques for cerclage are McDonald procedure and Shirodkar procedure. The McDonald procedure is easier to perform and remove. The bulk of data show no significant differences in pregnancy outcome between the two procedures (6, 9, 10).

McDonald cerclage -

* The procedure is begun by grasping the anterior and posterior lips of the cervix with one or two ring forceps
* A curved needle loaded with large caliber non-absorbable synthetic suture (at least number 1 or 2 braided or monofilament) is inserted at 12 o'clock, at least 2 cm above the external os.
* Four to six passes of a purse-string suture are taken circumferentially around the entire cervix as high as safely possible.
* The two ends of the suture are then tied securely and cut, leaving the ends long enough to grasp with a clamp when it is time to remove it (11).

During gestation, the female body undergoes hormonal, immunological, and metabolic changes to support fetal growth and development. There are noticeable changes in the microbiota at different body sites during pregnancy.

The human vaginal microbiota is a key component in the defense system against microbial and viral infections. The vaginal microbiome is dominated by many species including Lactobacillus and members of the Clostridiales, Bacteriodales, and Actinomycetales. Specifically, these lactic acid producing bacteria can create a barrier against pathogen invasion by maintaining a low pH (< 4.5) and by secreting metabolites that play an important role in inhibition of bacterial and viral infection in the urogenital tract.

The vaginal microbiome undergoes significant changes during pregnancy, including a significant decrease in overall diversity, increased stability and enrichment with Lactobacillus species (12). These correlate with a decrease in the vaginal pH and an increase in vaginal secretions. Vaginal microbial compositions were found to differ according to gestational age, while the communities at the later stages of pregnancy resembled those of the non-pregnant state. The dominant Lactobacillus species in pregnancy varies according to ethnic group. In women whose vaginal microbiota is not lactobacilli-dominated anti-bacterial defense mechanisms are reduced. The enhanced proliferation of pathogenic bacteria plus degradation of the cervical barrier increase bacterial passage into the endometrium and amniotic cavity and trigger preterm myometrial contractions (13).

About 2 million cervical cerclages are performed annually to prevent preterm birth. Two types of suture material are used for cerclage: monofilament or multifilament braided. Braided sutures are most frequently used, although no evidence exists to favor them over monofilament sutures. Birth outcomes in a retrospective cohort of 678 women receiving cervical cerclage in five UK university hospitals showed that braided cerclage was associated with increased intrauterine death (15% versus 5%; P = 0.0001) and preterm birth (28% versus 17%; P = 0.0006) compared to monofilament suture. A prospective study explored the vaginal microbiome in women at risk of preterm birth because of short cervical length (≤25 mm) who received braided (n = 25) or monofilament (n = 24) cerclage under comparable circumstances (14). Braided suture induced a persistent shift toward vaginal microbiome dysbiosis characterized by reduced Lactobacillus spp. and enrichment of pathobionts. Vaginal dysbiosis was associated with inflammatory cytokine and interstitial collagenase excretion into cervicovaginal fluid and premature cervical remodeling. Monofilament suture had comparatively minimal impact upon the vaginal microbiome and its interactions with the host. The shift of the human vaginal microbiome toward dysbiosis correlated with preterm birth (14).

ELIGIBILITY:
Inclusion Criteria:

* G- roup 1 - Pregnant women with a singleton gestation and cervical cerclage at 12-14 weeks of gestation due to obstetrical history characteristic of cervical insufficiency G- roup 2 - Pregnant women with a singleton gestation at 12-14 weeks of gestation without a history of cervical insufficiency
* Group 3 - Pregnant women treated with progesterone due to previous preterm labor without cerclage

Exclusion Criteria:

* A- cute cervical insufficiency P- roven or suspected chorioamnionitis P- remature rupture of membranes F- etal structural abnormality G- estation beyond 15 weeks A- ntibiotic usage in the past month P- robiotic use in the past month R- eported autoimmune disease or immunosuppressive disorder

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 100 (Estimated)
Dates: Start 2017-03-26 (Actual); Primary Completion 2020-01 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
vaginal microbiome distribution between the arms | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Maya Wolf, MD, Principal Investigator — Western Galilee Hospital
Locations (1):
- Galil Medical Center, Nahariya, Israel, Israel